CLINICAL TRIAL: NCT05583695
Title: Effects of Mindfulness-based Music Therapy on Emotional Regulation in Blind Elderly Women
Brief Title: Mindfulness-based Music Therapy in Blind Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RS-KHAB-2020-003
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Mindfulness; Music Therapy; Blind; Elderly; Mood

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mindfulness-based music therapy (Experimental)
  Interventions: Behavioral: mindfulness-based music therapy
- mindfulness-based therapy (Experimental)
  Interventions: Behavioral: mindfulness-based therapy
- routine care (Active Comparator)
  Interventions: Behavioral: routine care

INTERVENTIONS:
Behavioral: mindfulness-based music therapy — eight weekly sessions with a combination of both mindfulness and music therapy
  Arms: mindfulness-based music therapy
Behavioral: mindfulness-based therapy — eight weekly sessions of mindfulness
  Arms: mindfulness-based therapy
Behavioral: routine care — eight weekly sessions of routine care
  Arms: routine care

SUMMARY:
This trial aims to examine effects of mindfulness-based music therapy on mood regulation in blind elderly women.

ELIGIBILITY:
Inclusion Criteria:

* female
* blind with visual acuity (the best eye) of 20/400 or below
* aged 65 years or above
* cognitive intact, measured using Hong Kong Montreal Cognitive Assessment (6th version) with a score ≥ 12
* able to speak Cantonese

Exclusion Criteria:

* none

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | at baseline
  Difficulties in Emotion Regulation Scale is a 36-item measure assessing six emotion regulation dimensions: non-acceptance, goals, impulse, strategies, clarity, and awareness. The total score ranges from 36 to 180. Higher scores represent more difficultly in regulating emotions.
Difficulties in Emotion Regulation Scale (DERS) | In the 8th week from baseline
  Difficulties in Emotion Regulation Scale is a 36-item measure assessing six emotion regulation dimensions: non-acceptance, goals, impulse, strategies, clarity, and awareness. The total score ranges from 36 to 180. Higher scores represent more difficultly in regulating emotions.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales-21 (DASS-21) | at baseline
  Depression Anxiety Stress Scales-21 is a 21-item scale designed to assess depression, anxiety, and stress symptoms. It is divided into three subscales with each containing 7 items. Each subscale total score ranges from 0 to 21. Higher scores indicate more severe symptoms.
Depression Anxiety Stress Scales-21 (DASS-21) | In the 8th week from baseline
  Depression Anxiety Stress Scales-21 is a 21-item scale designed to assess depression, anxiety, and stress symptoms. It is divided into three subscales with each containing 7 items. Each subscale total score ranges from 0 to 21. Higher scores indicate more severe symptoms.
Geriatric Depression Scale (GDS) | at baseline
  Geriatric Depression Scale is a 30-item questionnaire asking how participants felt over the past week. The total score ranges from 0 to 30. Higher scores indicate more depressive symptoms.
Geriatric Depression Scale (GDS) | In the 8th week from baseline
  Geriatric Depression Scale is a 30-item questionnaire asking how participants felt over the past week. The total score ranges from 0 to 30. Higher scores indicate more depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Society for the Blind, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan SHW, Cheung MYC, Chiu ATS, Leung MHT, Kuo MCC, Yip DYC, Hui CCY, Kam SWI, Yeung K, Mui DSP, Wang SM, Yip CCK. Clinical effectiveness of mindfulness-based music therapy on improving emotional regulation in blind older women: A randomized controlled trial. Integr Med Res. 2023 Dec;12(4):100993. doi: 10.1016/j.imr.2023.100993. Epub 2023 Aug 26. PMID 37915438